CLINICAL TRIAL: NCT07384247
Title: Effect of Electrical Stimulation With Trigger Point Dry Needling on Pain and H-Reflex Muscle Activity
Brief Title: Trigger Point Dry Needling With and Without Electrical Stimulation in Healthy Subjects
Acronym: DN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, James Agostinucci, Associate Professor Sc.D., OTR/L, University of Rhode Island
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2122-042; IRB (Other: University of Rhode Island)
Record Dates: First submitted 2025-12-04; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: People With Identified Painful Trigger Points (Tp) Within the Soleus and Gastrocnemius Muscles Complex; Healthy Subjects or Volunteers
Keywords: dry needling; electrical stimulation; H-reflex; motor activity; pain threshold; trigger point
MeSH Terms: conditions — Motor Activity | interventions — Dry Needling; Electric Stimulation; Acupuncture Therapy; Electric Stimulation Therapy; Transcutaneous Electric Nerve Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy subjects who has identified painful trigger points within the soleus and gastrocnemius. (Experimental): This study was a randomized controlled trial. Forty volunteers, aged 18-55 were recruited, signed an informed consent and randomly placed in four equal groups: dry needling with simultaneous electrical stimulation, dry needling only, electrical stimulation only, and a Sham treatment.
  Interventions: Procedure: Dry needling with electrical stimulation; Procedure: Dry needling; Procedure: Electrical stimulation; Procedure: Sham

INTERVENTIONS:
Procedure: Dry needling with electrical stimulation — A dry needle inserted into the trigger point and left in the muscle for 10 min. Also, parameters of electrical stimulation were set at a frequency of 30 Hz and a pulse width of 0.6 ms, at an intensity that caused a small muscle contraction.
  Other Names: electrical dry needling
Procedure: Dry needling — A dry needle inserted into the trigger point and left in the muscle for 10 min. To ensure uniformity in conditions across all groups, a placebo electrical stimulation protocol was implemented, characterized by the initiation of electrical stimulation followed by its immediate cessation.
  Other Names: trigger point dry needling; acupuncture
Procedure: Electrical stimulation — Electrical stimulation setting is same as above dry needling with electrical stimulation group while the needle touch the skin to cause a prick over the muscle and were held there for 10 min.
  Other Names: electrotherapy; electrostimulation; electrical muscle stimulation; neuromuscular electrical stimulation; transcutaneous electrical nerve stimulation (TENS)
Procedure: Sham — The needle touches the skin to cause a prick over the muscle and were held there for 10 min (placebo dry needling) with placebo electrical stimulation which means initiating electrical stimulation but removing it instantaneously.
  Other Names: placebo

SUMMARY:
DN is one of the most commonly used physical therapy (PT) interventions for managing trigger points (Tp). Evidence suggests that DN was equally effective as other PT interventions, compared to no treatment or Sham-DN. Electrical stimulation (ES) is also a commonly used non-invasive method for pain management during PT. Recently, several studies suggested that combining DN with ES may be more effective in trigger point release than DN alone. The goal of this clinical trial was to determine the effects that trigger point dry needling with and without electrical stimulation had on pain threshold. It would also learn about the effect the trigger point dry needling has on muscle activity in people with identified painful trigger points within the soleus and gastrocnemius muscle complex. The main questions it aims to answer are:

* In terms of trigger point pain threshold, is DN combined with ES superior to DN alone, ES alone, or Sham treatment?
* In terms of muscle activity, is DN with ES superior to DN only, ES only or Sham treatment? Researchers will compare dry needling with electrical stimulation, dry needling only, electrical stimulation only and a Sham treatment to see these interventions affect pain threshold and muscle activity.

Participants will:

* Randomly assigned as one of the four groups
* Visit the clinic once for test
* Receive permission and conduct intervention according to protocol.

ELIGIBILITY:
Inclusion Criteria: healthy volunteers with at least 2 ≥ identifiable trigger points in soleus or gastrocnemius

Exclusion Criteria:

Age < 18 or > 55, able to communicate in English, no medical illness, or allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
To determine the effects that trigger point dry needling with and without electrical stimulation has on pain threshold | This was a single time point study. Pain threshold was assessed before (baseline) and at 10 and 30 mins post treatment.
  Primary outcome measure: when subjects perceived the intensity to be 50% of their maximum pain, based on a 1-10 analog pain scale.
  Participants held a switch with a button connected to a Bluetooth-enabled PS 850 Data Log (Biometrics Ltd., UK) data acquisition software system, where all pain recordings were analyzed and stored. The pain threshold was measured three times and averaged. We also checked visual analogue scale (VAS).

OTHER OUTCOMES:
To investigate the effects that trigger point dry needling with and without electrical stimulation has on the muscle activity (H-reflex) within the soleus and gastrocnemius muscles | This was a single time point study. Muscle activity was assessed before (baseline) and at 10 and 30 mins post treatment.
  Other outcome measure: Muscle activity was assessed using the H-reflex technique when the H-reflex amplitude was 15-25% of Mmax (H25%).
  Surface electrodes were used to stimulate the tibial nerve and record the H-reflex data. The H-reflex was elicited by a 2.5 cm monopolar stimulating ball electrode placed on the skin over the tibial nerve in the popliteal fossa.
  Ten Mmax responses were recorded. The electrical intensity was then lowered such that the H-reflex amplitude was 15-25% of Mmax (H25%). Ten H25% responses were recorded, and their averages served as the baseline data.

CONTACTS AND LOCATIONS:
Locations (1):
- Doctor of Physical Therapy, University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
This study was completed two years ago and received Institutional Review Board (IRB) approval; however, I require this approval for the submission of an original article.